CLINICAL TRIAL: NCT06680219
Title: A Single Centre, Double Blind, Placebo Controlled, Randomised Clinical Study Design in Healthy Subjects to Evaluate the Efficacy of a Digestive Health Supplement
Brief Title: Evaluation of the the Efficacy of a Digestive Health Supplement in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RIGSUP2C; RIGSUP2C (Other: PCR Corportation)
Record Dates: First submitted 2024-10-21; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects
Keywords: Nu Biome; abdominal discomfort logs; bloating

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo controlled, randomised 4-week home use study (Placebo Comparator): The sample is Crystal Light Raspberry Lemonade
  Placebo sample Usage instructions for all groups:
  2. Mix 3 scoops of powder (with scoop provided) with 8-12 oz of water. Enjoy once daily (8-12 oz of water is approximately 236-354 mL of water).
  Interventions: Dietary Supplement: Placebo
- Active comparator for randomised 4-week home use study (Active Comparator): ACTIVE - Nu Biome (Formula #: 95001996; Batch #: EV24931)
  Active sample Usage instructions for all groups:
  1. Mix 3 scoops of powder (with scoop provided) with 8-12 oz of water. Enjoy once daily (8-12 oz of water is approximately 236-354 mL of water).
  Interventions: Dietary Supplement: Active comparator

INTERVENTIONS:
Dietary Supplement: Placebo — Crystal Light Raspberry Lemonade: Mix 3 scoops of powder (with scoop provided) with 8-12 oz of water. Enjoy once daily (8-12 oz of water is approximately 236-354 mL of water).
  Arms: Placebo controlled, randomised 4-week home use study
Dietary Supplement: Active comparator — ACTIVE - Nu Biome (Formula #: 95001996; Batch #: EV24931): Mix 3 scoops of powder (with scoop provided) with 8-12 oz of water. Enjoy once daily.
  (8-12 oz of water is approximately 236-354 mL of water).
  Arms: Active comparator for randomised 4-week home use study

SUMMARY:
The objective of this study is to evaluate the efficacy of a digestive health supplement via waist circumference measurements, daily bowel habit and symptom logs, and self-perception questionnaires (SPQ) over 4 weeks.

To test for the following claims:

* Reduction of bloating after only one use.
* SPQ claims - to be determined by the sponsor.
* Improvement to a range of upper and lower gastrointestinal symptoms (heartburn, belching, bloating, nausea, vomiting, flatulence, intestinal cramps, urge to defecate, loose stool, and diarrhea)
* Clinically proven formulation
* Supports relief of bloating discomfort
* Supports quick and effective reduction in bloating related to food intake
* Study shows X% severity reduction in abdominal bloating
* Helps support a reduction in days experiencing bloating
* Supports a reduction in abdominal discomfort
* X% of participants reported a reduction in bloating during the study
* Supports a reduction in waist circumference, related to bloating

Please note that it is the responsibility of the sponsor to determine the testing and study designs required for submission to entities such as the Home Shopping Network, QVC, etc.

DETAILED DESCRIPTION:
Title: A single centre, double blind, placebo controlled, randomised clinical study design in healthy subjects to evaluate the efficacy of a digestive health supplement.

Study design: Single centre, placebo controlled, randomised 4-week home use study.

Test article: 1. ACTIVE - Nu Biome (Formula #: 95001996; Batch #: EV24931) 2. PLACEBO - Crystal Light Raspberry Lemonade

Duration of study: Approximately 4 weeks

Number of subjects: Enough subjects will be recruited onto the study to finish with 50 subjects overall across two (2) study groups:

Group 1: at least 20 subjects in the placebo group.

Group 2: at least 30 subjects in the active test article group.

Types of subjects: Healthy male and female subjects aged 20 - 60 years old including a range of ethnicities. Subjects must routinely experience gastrointestinal discomfort, specifically bloating.

Observations: Assessments for the randomised home use 4-week study consist of the following:

* Daily bowel habits log.
* Daily abdominal discomfort logs covering upper and lower gastrointestinal (GI) issues.
* Digestion-associated Quality of Life Questionnaire (DQLQ) at baseline, week 2, and week 4.
* Self-perception questionnaire for bloating at the 1st study visit (baseline and after 1 hour), at the 2nd study visit after 2 weeks of home use, and at the 3rd study visit after 4 weeks of home use (baseline and after 1 hour).
* Waist circumference measurements at the 1 st study visit (baseline and after 1 hour), at the 2nd study visit after 2 weeks of home use, and at the 3rd study visit after 4 weeks of home use (baseline and after 1 hour).
* Digital Photography of 20 subjects (10 from Group 1, 10 from Group 2) at the 1st study visit (baseline and after 1 hour), and at the 3rd study visit after 4 weeks of home use (baseline and after 1 hour).

ELIGIBILITY:
Inclusion Criteria

1. Healthy male and female subjects aged 20 - 60 years old including a range of ethnicities.
2. Subject routinely experiences gastrointestinal discomfort, specifically bloating.
3. Subject has signed a written Informed Consent.
4. Willing to use the test article as instructed following the directions for usage provided by the sponsor.
5. Willing to attend study visits 1 and 3 having fasted for 8 hours (only water allowed).
6. Willing to consume a test meal in conjunction with the supplement on study visits 1 and 3.
7. Willing to record daily logs of their bowel habits and abdominal discomfort.
8. Willing to attend all study visits.
9. Photography subjects: subjects undergoing clinical photography of the abdomen area are willing to wear the same clothing to visits 1 and 3 (or at least the same colour clothing).

Exclusion Criteria

1. Subject is pregnant, nursing, or planning to become pregnant.
2. Treatment or medication containing sympathomimetics, antihistamines or corticosteroids in the seven days prior to study start.
3. Known allergies or hypersensitivity to dietary supplements, similar materials, or their ingredients including, but not limited to, hazelnuts, peanuts and pomegranates (family Lythraceae).
4. Subject has allergies or sensitivity (other than bloating/indigestion issues/GI discomfort) to the ingredients of the test meal.
5. Insulin dependent diabetes.
6. Subjects with history of any gastrointestinal surgery, gastrointestinal illness which in the opinion of the Investigator would affect the digestive and absorption processes of the body (i.e., Gastric bypass, Gastroenteritis, Irritable Bowel Syndrome, Celiac Disease).
7. Medical condition that may affect study data or subject safety which in the opinion of the Investigator would compromise the safety of the subject or study results.
8. History of poor cooperation, non-compliance, or unreliability.
9. Investigator deems the subject an unsuitable candidate for the study.
10. Subject is currently participating in another clinical trial involving dietary supplements or similar materials.
11. Subject uses any prescription or over the counter (OTC) medication, vitamins, herbal products, antacids, mineral supplements and dietary supplements that target digestive issues and bloating within 4 weeks prior to the study start and through the end of study.
12. Chronic use of NSAIDs (e.g., Ibuprofen, Advil), or use of NSAIDs at one-week prior to each study Visit.
13. Subjects being treated with any known enzyme-altering drugs such as barbiturates, glucocorticoids, macrolides, antidepressants, neuroleptics, imidazole's, fluoroquinolones, calcium channel blockers, proton pump inhibitors, or H2-receptor antagonists, etc., within 30 days prior to screening or through the end of study.
14. Subjects with difficulty fasting or consuming standard meals or snacks.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Daily bowel habits log | 30 days
  Subjects in both arms will be asked to record their daily bowel habits in a diary using Bristol stool chart as a reference.
Daily abdominal discomfort assessment | 30 days
  Daily abdominal discomfort assessment will be recorded by subjects in a diary using Bristol Stool Chart as a reference on a scale of 0 to 10, with 0 (no discomfort) to 10 (worst discomfort).
Digestion-associated Quality of Life Questionnaire (DQLQ) assessment | 30 days
  Digestion-associated Quality of Life Questionnaire (DQLQ) will be assessed on a scale of 0% to 100% at baseline, week 2, and week 4, with 0% indicating no effect (never) on digestion-associated quality of life to 90%-100% (always effecting digestion-associated Quality of Life)
Self-perception questionnaire for assessment of bloating | 30 days
  Assessment of bloating using a self-perception questionnaire on a scale of None (no bloating) to very severe (severe bloating) will be conducted at the 1st study visit (baseline and after 1 hour), at the 2nd study visit after 2 weeks of home use, and at the 3rd study visit after 4 weeks of home use (baseline and after 1 hour).

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Drewitt, Principal Investigator — PCR Corp; Jamie Jarvis, Principal Investigator — PCR Corp
Locations (1):
- PCR Corp, Chelmsford, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No